CLINICAL TRIAL: NCT04588779
Title: Comparison of Graston and Manual Myofacial Release Technique in Patients With Piriformis Syndrome.
Brief Title: Graston vs Manual Myofascial Release Technique in Piriformis Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00689 Sonia Wali
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Piriformis Syndrome
Keywords: Graston technique; Myofascial release; Lower extremity functional scale; Piriformis syndrome
MeSH Terms: conditions — Piriformis Muscle Syndrome

STUDY DESIGN:
Intervention Model Description: Both groups were treated simultaneously with their specified treatment techniques within given duration.
Who Masked: Participant
Masking Description: Participants did not know which treatment techniques are given in the specified groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graston (Experimental): Ultrasound, Graston technique, piriformis stretching, home plan (hip abductor and extensor strengthening)
  Interventions: Other: Graston
- Manual myofascial release (Active Comparator): Ultrasound, Manual myofascial release, piriformis stretching, home plan (hip abductor and extensor strengthening)
  Interventions: Other: Manual myofascial release

INTERVENTIONS:
Other: Graston — Ultrasound for 10 mins/1 set/ (3 sessions/week), Graston for 5 mins/1 set/ (3 sessions/week), Piriformis stretching exercises/ 10 reps with 30 sec hold/ 1 set/(3 sessions/week), Hip abductor strengthening/10 reps/1 set/(3 weeks), Hip extensor strengthening/10 reps/1 set/(3 weeks),
  A total of 9 sessions for 3 weeks (3 sessions/week) were given each consisting of 20 mins.
  Arms: Graston
Other: Manual myofascial release — Ultrasound for 10 mins/1 set/ (3 sessions/week), Manual myofascial release for 5 mins/1 set/ (3 sessions/week), Piriformis stretching exercises/ 10 reps with 30 sec hold/ 1 set/(3 sessions/week), Hip abductor strengthening/10 reps/1 set/(3 weeks), Hip extensor strengthening/10 reps/1 set/(3 weeks),
  A total of 9 sessions for 3 weeks (3 sessions/week) were given each consisting of 20 mins.
  Arms: Manual myofascial release

SUMMARY:
The objective of our study is to compare the effects of Graston and manual myofascial release technique on pain, muscle length and functional status in patients with Piriformis syndrome.

DETAILED DESCRIPTION:
In 2019, a study was conducted to conclude the effectiveness of Passive stretching v/s Myofascial release in improving Piriformis flexibility in females. They reported that myofascial release was more valuable than passive stretching exercises in enhancing piriformis flexibility in patients with piriformis tightness.

According to another study in 2018, after a single treatment, compressive myofascial release showed more improvement in ankle dorsiflexion than Graston technique, in participants with decrease dorsiflexion range.

In 2016, a study reported the effects of the Graston technique and general exercise in patients with chronic low back pain. Graston group showed greater improvement in pain and range of motion in patients with chronic low back pain.

According to a study conducted in 2014, self-myofascial release was more effective than Graston technique in improving knee joint flexibility, hamstring, and quadriceps strength.

In 2011, a study evaluated the effectiveness of deep soft tissue mobilization techniques and stretching exercises in piriformis syndrome and found that the deep soft tissue mobilization techniques along with stretching exercises significantly improved the piriformis syndrome.

ELIGIBILITY:
Inclusion Criteria:•

* Pain more than 1 month.
* Piriformis syndrome diagnosed through screening test (FAIR test, Beatty test, Freiberg test, Sign of Pace)

Exclusion Criteria:

* Leg pain due to causes other than piriformis syndrome.
* Congenital spinal deformity.
* History of fracture.
* History of back or hip surgery.
* Any systemic illness like metastatic or infective disorders.

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — According to the feasibility of patients and examiner for assessment, only female patients were included in the study.
Enrollment: 30 (Actual)
Dates: Start 2020-01-11 (Actual); Primary Completion 2020-09-17 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 9th day
  Changes from baseline and after 1st session, Numeric pain rating scale is a scale from 0 to 10. 0 indicating no pain and 10 indicating worse pain.
Piriformis muscle length | 9th day
  Changes from baseline and after 1st session, in prone lying range of internal rotation is measured for piriformis muscle length
Lower extremity functional scale | 9th day
  Changes from baseline and after 1st session, lower extremity functional scale is used to measure the functional status of patients with piriformis syndrome.

SECONDARY OUTCOMES:
Straight leg raise | 9th day
  Changes from baseline and after 1st session, goniometer is used to measure the straight leg raise range.

CONTACTS AND LOCATIONS:
Overall Officials: Asghar Khan, Phd, Principal Investigator — Riphah International University
Locations (1):
- Federal government polyclinic hospital, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kukadia HA, Malshikare A, Palekar TJ. Effect of Passive Stretching v/s Myofascial Release in Improving Piriformis Flexibility in Females-A Comparative Study. Indian Journal of Physiotherapy and Occupational Therapy-An International Journal. 2019;13(4):57-61.
- [Background] Stanek J, Sullivan T, Davis S. Comparison of Compressive Myofascial Release and the Graston Technique for Improving Ankle-Dorsiflexion Range of Motion. J Athl Train. 2018 Feb;53(2):160-167. doi: 10.4085/1062-6050-386-16. Epub 2018 Jan 26. PMID 29373060
- [Background] Lee JH, Lee DK, Oh JS. The effect of Graston technique on the pain and range of motion in patients with chronic low back pain. J Phys Ther Sci. 2016 Jun;28(6):1852-5. doi: 10.1589/jpts.28.1852. Epub 2016 Jun 28. PMID 27390432
- [Background] Kim D-H, Ms T-HK, Jung D-Y, Weon J-H. Effects of the graston technique and self-myofascial release on the range of motion of a knee joint. Journal of Korean Society of Physical Medicine. 2014;9(4):455-63.
- [Background] Awan WA, Babur MN. EFFECTIVENESS OF DEEP FRICTION MASSAGE & STRETCHING EXERCISES IN PIRIFORMIS SYNDROME. IJCRB. 2011:378.